CLINICAL TRIAL: NCT01253590
Title: Feasibility of Remote Cardiac Monitoring of Post-Operative Cancer Patients Experiencing Atrial Fibrillation
Brief Title: Cardiac Monitoring of Post-Operative Cancer Patients Experiencing Atrial Fibrillation
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-213
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Post-Operative Cancer Patients Experiencing Atrial; Fibrillation
Keywords: atrial fibrillation; ECG monitor; Blood pressure device; Remote Cardiac Monitoring
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- post op cancer patients experiencing atrial fibrillation: This small study aims to assess the feasibility and acceptance of remote cardiac monitoring of postoperative cancer patients experiencing atrial fibrillation and will collect continuous data on heart beat over a period of 4-6 weeks upon discharge.
  Interventions: Behavioral: questionnaire about the use of ECG device

INTERVENTIONS:
Behavioral: questionnaire about the use of ECG device — Patients will be fitted with a continuous ECG monitor and blood pressure device. Data on every heart beat, including episodes of atrial fibrillation, for 4-6 weeks of continuous monitoring will be collected and transmitted wirelessly. Based on this information and blood pressure readings performed by patients in their home setting, clinicians can adjust oral coagulant dosage. Participants will attend 2 follow-up outpatient visits at the MSKCC outpatient cardiology practice upon the cardiologist's recommendation. Upon completion of the study, 4-6 weeks, a questionnaire will be sent via mail, including a pre-paid envelope, to participants to assess feasibility, acceptance, and overall experience with remote cardiac monitoring.
  Other Names: Upon obtaining written informed consent, a technician from Ocean Empire; Diagnostic & Monitoring Group will equip the participant with the ECG device and; demonstrate the use. This is standard practice at MSKCC for 24 hour holters; and we will be using the same company to equip patients with the ECG device.; Participants will also be equipped with a blood pressure device for use at; home during the 4-6 week period and the RN will demonstrate its use.

SUMMARY:
The purpose of this study is to assess whether it is possible and acceptable to monitor patients at a distance who experience a condition called atrial fibrillation after their cancer surgery. Some patients have no other clinical reason for staying in the hospital after cancer surgery except in order to control their heart rhythm. Being able to send these patients home earlier and monitor them at a distance from their home can be good for their quick recovery. Studies have shown greater quality of life and patient satisfaction when patients are monitored at a distance for conditions like atrial fibrillation, however cancer patients have not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Post-Operative cancer patients experiencing atrial fibrillation and otherwise clinically ready to be discharged.
* Must attend two outpatient visits at MSKCC's cardiology practice during the study period, as specified by the participant's Attending.
* Must be older than 21 years of age.

Exclusion Criteria:

* Non-English speaking patients

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two cardiology attending physicians, Dr. Michelle Johnson and Dr. Carol L. Chen, who are members of this research team, will identify post-operative patients whose primary attending has made a decision to discharge.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility and acceptance of continuous remote cardiac monitoring | 4 to 6 weeks
  In post-operative patients with respect to recurrence of post-operative atrial fibrillation upon discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Johnson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm